CLINICAL TRIAL: NCT02202980
Title: A Phase 2, Multicenter, Open-Label Study to Assess the Efficacy and Safety of Oral Regimens for the Treatment of Chronic HCV Infection
Brief Title: Efficacy and Safety of Oral Regimens for the Treatment of Chronic HCV Infection
Acronym: LEPTON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1468
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2017-11

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — ledipasvir, sofosbuvir drug combination; sofosbuvir-velpatasvir drug combination; voxilaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (15):
- LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1) (Experimental): Participants who previously received ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) plus ribavirin (RBV) for ≥ 12 weeks without achieving sustained virologic response at 12 weeks following treatment (SVR12) will receive LDV/SOF+RBV for 24 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF+RBV 12 Weeks (Cohort 1 Group 2) (Experimental): Participants who previously received a sofosbuvir-based regimen without achieving SVR12 were initially enrolled to receive LDV/SOF+RBV for 12 weeks (excluding participants who previously received LDV/SOF+RBV for ≥ 12 weeks). Participants who did not achieve sustained virologic response at 12 weeks were then moved to Cohort 1 Group 1.
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF 12 Weeks GT2 (Cohort 2 Group 1) (Experimental): Participants with genotype 2 (GT2) HCV infection will receive LDV/SOF FDC for 12 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF 8 Weeks GT2 (Cohort 2 Group 2) (Experimental): Participants with GT2 HCV infection will receive LDV/SOF FDC for 8 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF 12 Weeks GT1/GT2/GT4 (Cohort 3 Group 1) (Experimental): Participants with genotypes 1 (GT1), 2 (GT2), or 4 (GT4) HCV infection and extrahepatic manifestations of chronic HCV infection will receive LDV/SOF FDC for 12 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV 12 Weeks GT3 (Cohort 3 Group 2) (Experimental): Participants with genotype 3 (GT3) HCV infection and extrahepatic manifestations of chronic HCV infection will receive LDV/SOF FDC plus RBV for 12 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV
- SOF/VEL+VOX 6 Weeks GT1 (Cohort 4) (Experimental): Treatment-naive participants with GT1 HCV infection without cirrhosis will receive VOX only on Day 1 followed by sofosbuvir/velpatasvir (SOF/VEL) + voxilaprevir (VOX) for 6 weeks.
  Interventions: Drug: SOF/VEL; Drug: VOX
- SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1) (Experimental): Treatment-naive participants with GT1 HCV infection without cirrhosis will receive SOF/VEL+VOX for 4 weeks.
  Interventions: Drug: SOF/VEL; Drug: VOX
- SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2) (Experimental): Treatment-naive participants with GT1 HCV infection with cirrhosis will receive SOF/VEL+VOX for 6 weeks.
  Interventions: Drug: SOF/VEL; Drug: VOX
- SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3) (Experimental): Treatment-naive participants with GT3 HCV infection with cirrhosis will receive SOF/VEL+VOX for 6 weeks.
  Interventions: Drug: SOF/VEL; Drug: VOX
- SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4) (Experimental): Treatment-experienced participants with GT1 HCV infection with cirrhosis who were previously treated with pegylated interferon (Peg-IFN)+RBV will receive SOF/VEL+VOX for 6 weeks.
  Interventions: Drug: SOF/VEL; Drug: VOX
- SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5) (Experimental): Treatment-experienced participants with GT3 HCV infection with cirrhosis who were previously treated with Peg-IFN+RBV will receive SOF/VEL+VOX for 6 weeks.
  Interventions: Drug: SOF/VEL; Drug: VOX
- SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6) (Experimental): Treatment-experienced participants with GT1 HCV infection with or without cirrhosis who were previously treated with non-structural protein (NS3/4A) protease inhibitor (PI) will receive SOF/VEL+VOX for 6 weeks.
  Interventions: Drug: SOF/VEL; Drug: VOX
- SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7) (Experimental): Treatment-experienced participants with GT1 HCV infection with or without cirrhosis who were previously treated with direct-acting antivirals (DAA) will receive SOF/VEL+VOX for 6 weeks.
  Interventions: Drug: SOF/VEL; Drug: VOX
- SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8) (Experimental): Treatment-experienced participants with GT3 HCV infection with or without cirrhosis who were previously treated with DAA will receive SOF/VEL+VOX for 8 weeks.
  Interventions: Drug: SOF/VEL; Drug: VOX

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
  Arms: LDV/SOF 12 Weeks GT1/GT2/GT4 (Cohort 3 Group 1); LDV/SOF 12 Weeks GT2 (Cohort 2 Group 1); LDV/SOF 8 Weeks GT2 (Cohort 2 Group 2); LDV/SOF+RBV 12 Weeks (Cohort 1 Group 2); LDV/SOF+RBV 12 Weeks GT3 (Cohort 3 Group 2); LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1)
Drug: RBV — Tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: LDV/SOF+RBV 12 Weeks (Cohort 1 Group 2); LDV/SOF+RBV 12 Weeks GT3 (Cohort 3 Group 2); LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1)
Drug: SOF/VEL — 400/100 mg FDC tablet administered orally once daily
  Other Names: Epclusa®; GS-7977/GS-5816
  Arms: SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1); SOF/VEL+VOX 6 Weeks GT1 (Cohort 4); SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2); SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7); SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3); SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4); SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6); SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5); SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8)
Drug: VOX — 100 mg tablet administered orally once daily with food
  Other Names: GS-9857
  Arms: SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1); SOF/VEL+VOX 6 Weeks GT1 (Cohort 4); SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2); SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7); SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3); SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4); SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6); SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5); SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8)

SUMMARY:
This study will evaluate the antiviral efficacy, safety, and tolerability of combination therapy with oral regimens for the treatment of chronic hepatitis C virus (HCV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* Chronic HCV infection
* Cirrhosis determination (liver biopsy may be required)
* Screening laboratory values within specified limits
* Males and females of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
* Specific genotype, prior medical history, or concurrent disease as required by the specific study group

Key Exclusion Criteria:

* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol
* Pregnant or nursing female, or male with pregnant female partner
* Clinical hepatic decompensation (ie, ascites, encephalopathy or variceal hemorrhage)
* Use of any prohibited concomitant medications

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2016-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (2):
- New Zealand (2):
  - Auckland
  - Christchurch

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Gane EJ, Svarovskaia ES, Hyland RH, Stamm LM, Osinusi A, Brainard DM, Chodavarapu K, Miller MD, Mo H, Schwabe C. Resistance Analysis of Treatment-Naive and DAA-Experienced Genotype 1 Patients with and without Cirrhosis Who Received Short-Duration Treatment with Sofosbuvir/GS-5816+ GS-9857 [Poster 713]. J Hepatol 2015;62:563A
- [Result] Gane EJ, Schwabe C, Hyland RH, Yang Y, Svarovskaia E, Stamm LM, Brainard DM, McHutchison JG, Stedman CA. Efficacy of the Combination of Sofosbuvir, Velpatasvir, and the NS3/4A Protease Inhibitor GS-9857 in Treatment-Naive or Previously Treated Patients With Hepatitis C Virus Genotype 1 or 3 Infections. Gastroenterology. 2016 Sep;151(3):448-456.e1. doi: 10.1053/j.gastro.2016.05.021. Epub 2016 May 27. PMID 27240903
- [Result] Gane EJ, Hyland RH, Yang Y, Svarovskaia E, Stamm LM, Brainard DM, McHutchison JG, Stedman CAM. Efficacy of Ledipasvir Plus Sofosbuvir for 8 or 12 Weeks in Patients With Hepatitis C Virus Genotype 2 Infection. Gastroenterology. 2017 May;152(6):1366-1371. doi: 10.1053/j.gastro.2017.01.017. Epub 2017 Jan 27. PMID 28137593

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in New Zealand. The first participant was screened on 04 August 2014. The last study visit occurred on 09 May 2016.
Pre-assignment Details: 349 participants were screened.
Groups:
- LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1): Ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) + ribavirin (RBV) (1000 or 1200 mg daily based on weight) for 24 weeks in participants who previously received LDV/SOF+RBV for ≥ 12 weeks without achieving sustained virologic response at 12 weeks following treatment (SVR12)
- LDV/SOF 12 Weeks GT2 (Cohort 2 Group 1): LDV/SOF (90/400 mg) for 12 weeks in participants with genotype 2 HCV infection
- LDV/SOF 8 Weeks GT2 (Cohort 2 Group 2): LDV/SOF (90/400 mg) for 8 weeks in participants with genotype 2 HCV infection
- LDV/SOF 12 Weeks GT1/GT2/GT4 (Cohort 3 Group 1): LDV/SOF (90/400 mg) for 12 weeks in participants with genotypes 1, 2, or 4 HCV infection and extrahepatic manifestations of chronic HCV infection
- LDV/SOF 12 Weeks GT3 (Cohort 3 Group 2): LDV/SOF (90/400 mg) + RBV (1000 or 1200 mg daily based on weight) for 12 weeks in participants with genotype 3 HCV infection and extrahepatic manifestations of chronic HCV infection
- SOF/VEL+VOX 6 Weeks GT1 (Cohort 4): Voxilaprevir (VOX) 100 mg with food on Day 1, followed by sofosbuvir/velpatasvir (SOF/VEL) (400/100 mg) + VOX 100 mg once daily with food for 6 weeks in treatment-naive participants with genotype 1 HCV infection without cirrhosis
- SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1): SOF/VEL (400/100 mg) + VOX 100 mg once daily with food for 4 weeks in treatment-naive participants with genotype 1 HCV infection without cirrhosis
- SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2): SOF/VEL (400/100 mg) + VOX 100 mg once daily with food for 6 weeks in treatment-naive participants with genotype 1 HCV infection with cirrhosis
- SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3): SOF/VEL (400/100 mg) + VOX 100 mg once daily with food for 6 weeks in treatment-naive participants with genotype 3 HCV infection with cirrhosis
- SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4): SOF/VEL (400/100 mg) + VOX 100 mg once daily with food for 8 weeks in treatment-experienced participants with genotype 1 HCV infection with cirrhosis
- SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5): SOF/VEL (400/100 mg) + VOX 100 mg once daily with food for 8 weeks in treatment-experienced participants with genotype 3 HCV infection with cirrhosis
- SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6): SOF/VEL (400/100 mg) + VOX 100 mg once daily with food for 8 weeks in nonstructural protein (NS3/4A) protease inhibitor (PI)-treatment-experienced participants with genotype 1 HCV infection with or without cirrhosis
- SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7): SOF/VEL (400/100 mg) + VOX 100 mg once daily with food for 6 weeks in direct-acting antiviral (DAA)-treatment-experienced participants with genotype 1 HCV infection with or without cirrhosis
- SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8): SOF/VEL (400/100 mg) + VOX 100 mg once daily with food for 8 weeks in DAA-treatment-experienced participants with genotype 3 HCV infection with or without cirrhosis
Period: Overall Study
Arm/Group | LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1) | LDV/SOF 12 Weeks GT2 (Cohort 2 Group 1) | LDV/SOF 8 Weeks GT2 (Cohort 2 Group 2) | LDV/SOF 12 Weeks GT1/GT2/GT4 (Cohort 3 Group 1) | LDV/SOF 12 Weeks GT3 (Cohort 3 Group 2) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 4) | SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2) | SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8)
Started | 14 | 26 | 27 | 32 | 13 | 15 | 15 | 15 | 18 | 17 | 19 | 28 | 30 | 4
Completed | 13 | 24 | 17 | 28 | 7 | 14 | 4 | 12 | 14 | 17 | 19 | 25 | 19 | 4
Not Completed | 1 | 2 | 10 | 4 | 6 | 1 | 11 | 3 | 4 | 0 | 0 | 3 | 11 | 0
Not completed — Lack of Efficacy | 1 | 0 | 7 | 0 | 3 | 1 | 11 | 2 | 2 | 0 | 0 | 3 | 10 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrew Consent | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were enrolled into the study and received at least 1 dose of study drug
Groups:
- LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1): LDV/SOF (90/400 mg) + RBV (1000 or 1200 mg daily based on weight) for 24 weeks in participants who previously received LDV/SOF+RBV for ≥ 12 weeks without achieving SVR12
- SOF/VEL+VOX 6 Weeks GT1 (Cohort 4): VOX 100 mg with food on Day 1, followed by SOF/VEL (400/100 mg) + VOX 100 mg once daily with food for 6 weeks in treatment-naive participants with genotype 1 HCV infection without cirrhosis
- SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6): SOF/VEL (400/100 mg) + VOX 100 mg once daily with food for 8 weeks in NS3/4A PI-treatment-experienced participants with genotype 1 HCV infection with or without cirrhosis
- SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7): SOF/VEL (400/100 mg) + VOX 100 mg once daily with food for 6 weeks in DAA-treatment-experienced participants with genotype 1 HCV infection with or without cirrhosis
- Total: Total of all reporting groups
Arm/Group | LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1) | LDV/SOF 12 Weeks GT2 (Cohort 2 Group 1) | LDV/SOF 8 Weeks GT2 (Cohort 2 Group 2) | LDV/SOF 12 Weeks GT1/GT2/GT4 (Cohort 3 Group 1) | LDV/SOF 12 Weeks GT3 (Cohort 3 Group 2) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 4) | SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2) | SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8) | Total
Number analyzed (Participants) | 14 | 26 | 27 | 32 | 13 | 15 | 15 | 15 | 18 | 17 | 19 | 28 | 30 | 4 | 273
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 24 | 25 | 29 | 13 | 13 | 15 | 14 | 18 | 16 | 18 | 26 | 29 | 4 | 257
  >=65 years | 1 | 2 | 2 | 3 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 8 | 12 | 1 | 8 | 6 | 4 | 8 | 3 | 4 | 9 | 6 | 0 | 82
  Male | 10 | 17 | 19 | 20 | 12 | 7 | 9 | 11 | 10 | 14 | 15 | 19 | 24 | 4 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 14 | 26 | 27 | 32 | 13 | 15 | 14 | 15 | 18 | 17 | 19 | 28 | 30 | 4 | 272
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 24 | 21 | 26 | 12 | 14 | 12 | 14 | 12 | 16 | 18 | 24 | 27 | 3 | 233
  Asian | 2 | 2 | 5 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 1 | 2 | 0 | 15
  Other | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 9
HCV genotype [Count of Participants; unit: Participants]
  Genotype 1a | 1 | 0 | 0 | 28 | 0 | 11 | 11 | 14 | 0 | 15 | 0 | 24 | 23 | 0 | 127
  Genotype 1b | 0 | 0 | 0 | 3 | 0 | 4 | 4 | 1 | 0 | 2 | 0 | 4 | 7 | 0 | 25
  Genotype 2 | 7 | 2 | 27 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36
  Genotype 2a or 2c | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Genotype 2b | 0 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  Genotype 3 | 2 | 0 | 0 | 0 | 12 | 0 | 0 | 0 | 17 | 0 | 19 | 0 | 0 | 4 | 54
  Genotype 3a | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Genotype 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Indeterminate | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Cirrhosis Status [Count of Participants; unit: Participants]
  Yes | 4 | 2 | 0 | 9 | 10 | 0 | 0 | 15 | 18 | 17 | 19 | 11 | 5 | 2 | 112
  No | 10 | 24 | 27 | 23 | 3 | 15 | 15 | 0 | 0 | 0 | 0 | 17 | 25 | 2 | 161
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 7 | 10 | 14 | 6 | 4 | 5 | 5 | 8 | 10 | 6 | 8 | 4 | 6 | 3 | 96
    CT | 7 | 15 | 10 | 18 | 6 | 8 | 10 | 7 | 6 | 9 | 9 | 21 | 18 | 1 | 145
    TT | 0 | 1 | 3 | 7 | 3 | 2 | 0 | 0 | 2 | 2 | 2 | 3 | 6 | 0 | 31
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 1 | 11 | 5 | 8 | 4 | 5 | 4 | 4 | 5 | 3 | 3 | 10 | 5 | 0 | 68
  ≥ 800,000 IU/mL | 13 | 15 | 22 | 24 | 9 | 10 | 11 | 11 | 13 | 14 | 16 | 18 | 25 | 4 | 205
Prior HCV Treatment [Count of Participants; unit: Participants]
  Treatment-Naive | 0 | 21 | 20 | 17 | 3 | 15 | 15 | 15 | 18 | 0 | 0 | 0 | 0 | 0 | 124
  Treatment-Experienced | 14 | 5 | 7 | 15 | 10 | 0 | 0 | 0 | 0 | 17 | 19 | 28 | 30 | 4 | 149

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were enrolled into the study and received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1) | LDV/SOF 12 Weeks GT2 (Cohort 2 Group 1) | LDV/SOF 8 Weeks GT2 (Cohort 2 Group 2) | LDV/SOF 12 Weeks GT1/GT2/GT4 (Cohort 3 Group 1) | LDV/SOF 12 Weeks GT3 (Cohort 3 Group 2) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 4) | SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2) | SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8)
Number analyzed (Participants) | 14 | 26 | 27 | 32 | 13 | 15 | 15 | 15 | 18 | 17 | 19 | 28 | 30 | 4
percentage of participants | 92.9 [66.1 to 99.8] | 96.2 [80.4 to 99.9] | 74.1 [53.7 to 88.9] | 100.0 [89.1 to 100.0] | 76.9 [46.2 to 95.0] | 93.3 [68.1 to 99.8] | 26.7 [7.8 to 55.1] | 86.7 [59.5 to 98.3] | 83.3 [58.6 to 96.4] | 100.0 [80.5 to 100.0] | 100.0 [82.4 to 100.0] | 89.3 [71.8 to 97.7] | 66.7 [47.2 to 82.7] | 100.0 [39.8 to 100.0]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set: participants who were enrolled into the study and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1) | LDV/SOF 12 Weeks GT2 (Cohort 2 Group 1) | LDV/SOF 8 Weeks GT2 (Cohort 2 Group 2) | LDV/SOF 12 Weeks GT1/GT2/GT4 (Cohort 3 Group 1) | LDV/SOF 12 Weeks GT3 (Cohort 3 Group 2) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 4) | SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2) | SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8)
Number analyzed (Participants) | 14 | 26 | 27 | 32 | 13 | 15 | 15 | 15 | 18 | 17 | 19 | 28 | 30 | 4
percentage of participants | 7.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set: participants who were enrolled into the study and received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1) | LDV/SOF 12 Weeks GT2 (Cohort 2 Group 1) | LDV/SOF 8 Weeks GT2 (Cohort 2 Group 2) | LDV/SOF 12 Weeks GT1/GT2/GT4 (Cohort 3 Group 1) | LDV/SOF 12 Weeks GT3 (Cohort 3 Group 2) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 4) | SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2) | SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8)
Number analyzed (Participants) | 14 | 26 | 27 | 32 | 13 | 15 | 15 | 15 | 18 | 17 | 19 | 28 | 30 | 4
percentage of participants
  SVR4 | 92.9 [66.1 to 99.8] | 96.2 [80.4 to 99.9] | 81.5 [61.9 to 93.7] | 100.0 [89.1 to 100.0] | 76.9 [46.2 to 95.0] | 100.0 [78.2 to 100.0] | 73.3 [44.9 to 92.2] | 86.7 [59.5 to 98.3] | 88.9 [65.3 to 98.6] | 100.0 [80.5 to 100.0] | 100.0 [82.4 to 100.0] | 92.9 [76.5 to 99.1] | 86.7 [69.3 to 96.2] | 100.0 [39.8 to 100.0]
  SVR24 | 92.9 [66.1 to 99.8] | 96.2 [80.4 to 99.9] | 74.1 [53.7 to 88.9] | 100.0 [89.1 to 100.0] | 76.9 [46.2 to 95.0] | 93.3 [68.1 to 99.8] | 20.0 [4.3 to 48.1] | 86.7 [59.5 to 98.3] | 83.3 [58.6 to 96.4] | 100.0 [80.5 to 100.0] | 100.0 [82.4 to 100.0] | 89.3 [71.8 to 97.7] | 66.7 [47.2 to 82.7] | 100.0 [39.8 to 100.0]

4. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set: participants who were enrolled into the study and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1) | LDV/SOF 12 Weeks GT2 (Cohort 2 Group 1) | LDV/SOF 8 Weeks GT2 (Cohort 2 Group 2) | LDV/SOF 12 Weeks GT1/GT2/GT4 (Cohort 3 Group 1) | LDV/SOF 12 Weeks GT3 (Cohort 3 Group 2) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 4) | SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2) | SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8)
Number analyzed (Participants) | 14 | 26 | 27 | 32 | 13 | 15 | 15 | 15 | 18 | 17 | 19 | 28 | 30 | 4
percentage of participants | 7.1 | 0 | 22.2 | 0 | 23.1 | 6.7 | 73.3 | 13.3 | 11.1 | 0 | 0 | 10.7 | 30.0 | 0

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ While on Treatment by Study Visit
Time Frame: Weeks 1, 2, 4, 6, 8, 12, 16, 20, and 24 (depending on treatment duration; Week 6 data was not collected for Cohorts 1-3)
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1) | LDV/SOF 12 Weeks GT2 (Cohort 2 Group 1) | LDV/SOF 8 Weeks GT2 (Cohort 2 Group 2) | LDV/SOF 12 Weeks GT1/GT2/GT4 (Cohort 3 Group 1) | LDV/SOF 12 Weeks GT3 (Cohort 3 Group 2) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 4) | SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2) | SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8)
Number analyzed (Participants) | 14 | 25 | 27 | 32 | 13 | 15 | 15 | 15 | 18 | 17 | 19 | 28 | 30 | 4
percentage of participants
  Week 1 | 7.1 | 28.0 | 7.4 | 9.4 | 7.7 | 26.7 | 26.7 | 26.7 | 16.7 | 5.9 | 5.3 | 7.1 | 13.3 | 0
  Week 2 | 64.3 | 60.0 | 40.7 | 53.1 | 7.7 | 66.7 | 53.3 | 66.7 | 88.9 | 41.2 | 42.1 | 60.7 | 43.3 | 25.0
  Week 4 | 100.0 | 92.0 | 92.6 | 87.5 | 84.6 | 100.0 | 100.0 | 100.0 | 100.0 | 76.5 | 84.2 | 85.7 | 93.3 | 100.0
  Week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 15 | 0 | 15 | 18 | 17 | 19 | 28 | 30 | 4
  Week 6 |  |  |  |  |  | 100.0 |  | 100.0 | 100.0 | 100.0 | 94.7 | 96.4 | 96.7 | 100.0
  Week 8: number analyzed (Participants) | 14 | 25 | 27 | 32 | 13 | 0 | 0 | 0 | 0 | 17 | 19 | 28 | 0 | 4
  Week 8 | 100.0 | 100.0 | 96.3 | 100.0 | 100.0 |  |  |  |  | 100.0 | 100.0 | 100.0 |  | 100.0
  Week 12: number analyzed (Participants) | 14 | 25 | 0 | 32 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 | 100.0 | 100.0 |  | 100.0 | 100.0 |  |  |  |  |  |  |  |  |
  Week 16: number analyzed (Participants) | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16 | 92.9 |  |  |  |  |  |  |  |  |  |  |  |  |
  Week 20: number analyzed (Participants) | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 20 | 92.9 |  |  |  |  |  |  |  |  |  |  |  |  |
  Week 24: number analyzed (Participants) | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 24 | 100.0 |  |  |  |  |  |  |  |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set: participants who were enrolled into the study and received at least 1 dose of study drug
Arm/Group | LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1) | LDV/SOF 12 Weeks GT2 (Cohort 2 Group 1) | LDV/SOF 8 Weeks GT2 (Cohort 2 Group 2) | LDV/SOF 12 Weeks GT1/GT2/GT4 (Cohort 3 Group 1) | LDV/SOF 12 Weeks GT3 (Cohort 3 Group 2) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 4) | SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2) | SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/26 | 0/27 | 0/32 | 0/13 | 0/15 | 0/15 | 0/15 | 0/18 | 0/17 | 0/19 | 0/28 | 0/30 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/14 | 1/26 | 2/27 | 3/32 | 2/13 | 0/15 | 0/15 | 0/15 | 0/18 | 0/17 | 2/19 | 1/28 | 0/30 | 0/4
Other Adverse Events (participants affected / at risk) | 12/14 | 15/26 | 21/27 | 24/32 | 11/13 | 12/15 | 13/15 | 10/15 | 15/18 | 15/17 | 14/19 | 21/28 | 23/30 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1) (N=14) | LDV/SOF 12 Weeks GT2 (Cohort 2 Group 1) (N=26) | LDV/SOF 8 Weeks GT2 (Cohort 2 Group 2) (N=27) | LDV/SOF 12 Weeks GT1/GT2/GT4 (Cohort 3 Group 1) (N=32) | LDV/SOF 12 Weeks GT3 (Cohort 3 Group 2) (N=13) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 4) (N=15) | SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1) (N=15) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2) (N=15) | SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3) (N=18) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4) (N=17) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5) (N=19) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6) (N=28) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7) (N=30) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8) (N=4)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF+RBV 24 Weeks (Cohort 1 Group 1) (N=14) | LDV/SOF 12 Weeks GT2 (Cohort 2 Group 1) (N=26) | LDV/SOF 8 Weeks GT2 (Cohort 2 Group 2) (N=27) | LDV/SOF 12 Weeks GT1/GT2/GT4 (Cohort 3 Group 1) (N=32) | LDV/SOF 12 Weeks GT3 (Cohort 3 Group 2) (N=13) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 4) (N=15) | SOF/VEL+VOX 4 Weeks GT1 (Cohort 5 Group 1) (N=15) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 2) (N=15) | SOF/VEL+VOX 6 Weeks GT3 (Cohort 5 Group 3) (N=18) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 4) (N=17) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 5) (N=19) | SOF/VEL+VOX 8 Weeks GT1 (Cohort 5 Group 6) (N=28) | SOF/VEL+VOX 6 Weeks GT1 (Cohort 5 Group 7) (N=30) | SOF/VEL+VOX 8 Weeks GT3 (Cohort 5 Group 8) (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 3 | 2 | 0 | 4 | 1 | 0 | 6 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 5 | 5 | 1 | 5 | 5 | 3 | 3 | 1 | 7 | 3 | 5 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 1 | 1 | 1 | 0 | 2 | 1 | 3 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 6 | 5 | 4 | 2 | 5 | 2 | 2 | 3 | 3 | 2 | 7 | 3 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 0 | 7 | 1 | 0 | 2 | 0 | 4 | 0 | 1 | 4 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 6 | 7 | 6 | 1 | 6 | 2 | 4 | 6 | 3 | 4 | 5 | 6 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Migraine without aura (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Irritability (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years